CLINICAL TRIAL: NCT06796907
Title: A Phase I/II Randomized Multi-Cohort Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Activity of GSK5733584 in Combination With Anti-Cancer Agents in Participants With Advanced Solid Tumors
Brief Title: A Study of GSK5733584 in Combination With Anti-cancer Therapies for Advanced Solid Tumors
Acronym: BEHOLD-2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 223559; 2024-517147-31-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Tumours, Gynecological
Keywords: Solid Tumors; GSK5733584; BEHOLD-2
MeSH Terms: conditions — Neoplasms | interventions — dostarlimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Module 1 (GSK5733584 +/- Dostarlimab) Endometrial Cancer (Experimental)
  Interventions: Drug: GSK5733584; Drug: Dostarlimab
- Module 2 (GSK5733584 +/- Bevacizumab) Ovarian Cancer (Experimental)
  Interventions: Drug: GSK5733584; Drug: Bevacizumab
- Module 3 (GSK5733584 + Anticancer therapy 3 +/- Dostarlimab or Bevacizumab) (Experimental)
  Interventions: Drug: GSK5733584; Drug: Dostarlimab; Drug: Bevacizumab; Drug: Anticancer therapy 3
- Module 4 (GSK5733584 + Anticancer therapy 4 +/- Dostarlimab or Bevacizumab) (Experimental)
  Interventions: Drug: GSK5733584; Drug: Dostarlimab; Drug: Bevacizumab; Drug: Anticancer therapy 4

INTERVENTIONS:
Drug: GSK5733584 — GSK5733584 will be administered intravenously (IV).
Drug: Dostarlimab — Dostarlimab will be administered IV.
  Arms: Module 1 (GSK5733584 +/- Dostarlimab) Endometrial Cancer; Module 3 (GSK5733584 + Anticancer therapy 3 +/- Dostarlimab or Bevacizumab); Module 4 (GSK5733584 + Anticancer therapy 4 +/- Dostarlimab or Bevacizumab)
Drug: Bevacizumab — Bevacizumab will be administered IV.
  Arms: Module 2 (GSK5733584 +/- Bevacizumab) Ovarian Cancer; Module 3 (GSK5733584 + Anticancer therapy 3 +/- Dostarlimab or Bevacizumab); Module 4 (GSK5733584 + Anticancer therapy 4 +/- Dostarlimab or Bevacizumab)
Drug: Anticancer therapy 3 — Anticancer therapy 3 will be administered IV.
  Arms: Module 3 (GSK5733584 + Anticancer therapy 3 +/- Dostarlimab or Bevacizumab)
Drug: Anticancer therapy 4 — Anticancer therapy 4 will be administered IV.
  Arms: Module 4 (GSK5733584 + Anticancer therapy 4 +/- Dostarlimab or Bevacizumab)

SUMMARY:
Advanced solid tumors are cancers that have spread to other parts of the body. While many treatments exist, most people become resistant to them, and the cancer returns. Researchers are developing new treatments that combine different medicines for those who do not respond to single medicine. This study is looking at how safe and tolerable GSK5733584 is, how the body handles it, and how well it works when used with other cancer medicines. The study will include participants with advanced solid tumors who have either not responded to standard treatments or cannot tolerate them or have no available effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age inclusive or older, at the time of signing the informed consent, or the legal age of consent in the jurisdiction in which the study is taking place.
* Participant capable of giving signed informed consent including compliance with the requirements and restrictions listed in the Informed consent form (ICF) and in this protocol.
* Participants with pathologically confirmed advanced solid tumor specific for study arms (key local diagnostic molecular and/or immunophenotyping testing results/tumor cell phenotype results for confirmed diagnosis should be provided) with no more than 4 lines of prior systemic therapies. Please note:

  1. Adjuvant +/- neoadjuvant considered one line of therapy
  2. Maintenance therapy will be considered as part of the preceding line of therapy (i.e., not counted independently)
  3. Unplanned addition or switching to a new drug in a different class is considered a separate line of therapy. If an agent in a regimen is switched to another agent in the same class due to toxicity or intolerance (e.g. hypersensitivity reaction) this is considered part of the same line (i.e. not counted independently).
* Requirements for tumor tissue samples: Archival or fresh tumor tissue is required for retrospective central assessment of B7H4 expression by immunohistochemistry (IHC) and other biomarker analysis. The archival tumor tissue should be from the most recent procedure (ideally obtained after the last anti-cancer treatment). If an archival tissue is not available a new biopsy should be performed, and the newly obtained tissue provided.
* Participants have at least one target lesion as assessed per RECIST 1.1. A target lesion is defined as a measurable lesion that has not undergone locoregional treatment such as irradiation or that has unequivocal progression following locoregional treatment, with the longest diameter of ≥ 10 millimeter (mm) at Baseline (for lymph node lesions, the short axis should be ≥ 15 mm).
* Participants have a life expectancy of at least 12 weeks per investigator assessment based on disease burden and extent of supportive care needed.

Inclusion criteria of participants under arm Module 1 (GSK5733584 +/- Dostarlimab) Endometrial Cancer Part A:

a. Participants with histologically documented, advanced (metastatic and/or unresectable) or recurrent endometrial cancer who have failed in adequate standard treatments, do not have effective standard treatment or are intolerant to standard of care, and who are not candidates for further curative external radiotherapy or brachytherapy.

Inclusion criteria of participants under arm Module 1 (GSK5733584 +/- Dostarlimab) Endometrial Cancer Part B:

1. Diagnosis of endometrial cancer with confirmed mismatch repair proficient (MMRp) or microsatellites stable (MSS) tumor status by local test.
2. Participants who have progressed on or are intolerant to at least 1 line of standard prior systemic therapy (including neoadjuvant or adjuvant as prior line), and who are not candidates for curative external radiotherapy or brachytherapy. Maintenance therapy will be considered part of the preceding line of therapy (i.e, not counted independently).
3. Participants naïve to anti-programmed death protein 1 and/or programmed death ligand 1 (PD[L]-1) anti-cancer therapy.

Inclusion criteria of participants under arm Module 2 (GSK5733584 +/- Bevacizumab) Ovarian Cancer Part A:

a. Participants with histologically or cytologically confirmed advanced epithelial ovarian cancer/fallopian tube/peritoneal cancer (any epithelial histology - mucinous, clear cell, carcinosarcoma, high/low grade serous, endometrioid) who have failed in adequate standard treatments, do not have effective standard treatment or are intolerant to standard of care.

Inclusion criteria of participants under arm Module 2 (GSK5733584 +/- Bevacizumab) Ovarian Cancer Part B:

1. Participants whose advanced ovarian cancer/fallopian tube/peritoneal cancer has relapsed more than 6 months from the last dose of platinum before enrollment, i.e., platinum sensitive.
2. Participants who have progressed on or are intolerant to at least 1 line of standard prior lines of chemotherapy and are not candidates for second cytoreductive surgery.

   * Participants willing to use adequate contraception.
   * Male participants:

     * Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 6 months after the last dose of study intervention for Arms 1 to 3 and 11 Months after the last dose of study intervention for Arm 4:
     * Refrain from donating sperm.
   * Female participants:

A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

* Is a Woman of non-childbearing potential (WONCBP) OR
* Is a Woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention

  * Has an ECOG performance status of 0 to 1.
  * Participants with normal organ and bone marrow function

Exclusion Criteria:

* Has a second malignancy (except disease under study) that has progressed or required active treatment within the past 24 months except for basal cell or squamous cell carcinomas of the skin or in-situ carcinomas [e.g., breast, cervix, bladder] that have been resected with no evidence of metastatic disease.
* Has any history of prior allogenic or autologous bone marrow transplant or other solid organ transplant.
* Has known sensitivity to study intervention components, GSK5733584 (antibody-drug conjugate, antibody, free cytotoxin GSK5757810A) and combination partner, or its excipients or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
* Has any following cardiological examination abnormality:

  1. history in prior year of clinically significant or uncontrolled cardiac disease, acute myocardial infarction, or clinically significant arrhythmia not controlled by standard of care therapy.
  2. Corrected QT Interval (QTcF) >450 millisecond (msec) or QTcF >480 msec for participants with bundle branch block
* Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis.
* Has a history of autoimmune disease that has required systemic treatments in the 2 years prior to screening (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy is not considered a form of systemic therapy (e.g., thyroid hormone for autoimmune thyroiditis or insulin is not exclusionary).
* Clinically significant bleeding symptoms, significant bleeding tendency, or bleeding tumors within 1 month prior to the first dose of study treatment.
* Serious or poorly controlled hypertension, including history of hypertensive crisis, hypertensive encephalopathy; adjustment of antihypertensive medications due to poor blood pressure control within 2 weeks prior to the first dose of study treatment; systolic blood pressure ≥ 160 millimeter of mercury (mmHg) or diastolic blood pressure ≥ 100 mmHg during screening period.
* Has any active renal condition (e.g., infection, requirement for dialysis, or any other active significant renal condition or dehydrated condition that could affect the participant's safety).
* Participants with known history of Human immunodeficiency virus (HIV).
* Has an Alanine transaminase (ALT) value >2.5x Upper Limit of Normal (ULN) and for participants with documented liver metastases/tumor infiltration has an ALT value >5x ULN.
* Has a total bilirubin value >1.5x ULN.
* Has received treatment with any cytotoxic chemotherapy drugs or other anti-tumor drugs (including endocrine therapy, molecular targeted therapy, immunotherapy, biotherapy, and investigational drug) within 30 days or 5 half-lives, whichever is shorter of a medicinal product prior to the first dose of study drug; or need to continue these drugs during the study.
* Use of strong or moderate inhibitors or inducers of CYP3A4, CYP2D6 and inhibitors or inducers of P-gp, and breast cancer resistance protein (BCRP) within 14 days prior to the first dose of study drug; or in need of continuing treatment with these drugs during the study.
* Have received locoregional radiation therapy within 2 weeks prior to the first dose of study drug; more than 30% of bone marrow irradiation or wide-field radiation therapy within 4 weeks prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2028-04-05 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of participants with dose limiting toxicities (DLTs) | Approximately 7 months
Part A: Number of participants with adverse events (AEs), immune-mediated adverse events (imAEs), adverse events of special interest (AESI), serious adverse events (SAEs) by Severity | Up to approximately 22 months
Part A: Number of participants with adverse events (AEs), immune-mediated adverse events (imAEs), adverse events of special interest (AESI), serious adverse events (SAEs) by Frequency | Up to approximately 22 months
Part B: Confirmed Objective Response Rate (ORR) | Up to approximately 37 months
  ORR is defined as the percentage of participants with a best overall confirmed (BOR) of Partial Response (PR) or better per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
Part A: Confirmed Objective Response Rate (ORR) | Up to approximately 22 months
  ORR is defined as the percentage of participants with a best overall confirmed (BOR) of PR or better per RECIST 1.1.
Parts A and B: Duration of response (DoR) | Up to approximately 37 months
  DoR is defined as the time from date of first documented evidence of PR or better to the date of disease progression or death due to any cause.
Parts A and B: Progression-free survival (PFS) | Up to approximately 37 months
  PFS is defined as time from the date of randomization (Part B) / first dose of study intervention (Part A or B if single arm) to the date of disease progression according to investigator assessment or death due to any cause, whichever occurs first.
Part B: Overall Survival (OS) | Up to approximately 37 months
  OS is defined as the time from randomization (or date of first dose if single arm) to the date of death due to any cause.
Parts A and B: Maximum observed concentration (Cmax) of GSK5733584 | Up to approximately 37 months
Parts A and B: Time to reach Cmax (tmax) of GSK5733584 | Up to approximately 37 months
Parts A and B: Trough concentration (Ctrough) of GSK5733584 | Up to approximately 37 months
Parts A and B: Area under the concentration-time curve (AUC) of GSK5733584 | Up to approximately 37 months
Parts A and B: Number of participants with Anti-drug antibodies (ADA) | Up to approximately 37 months
Parts A and B: Number of participants with neutralizing antibody (nAb) | Up to approximately 37 months
Parts A and B: Titers of ADA to GSK5733584 | Up to approximately 37 months
Parts A and B: Number of Participants with Clinically Significant Changes in Vital Signs, Laboratory parameters, and Electrocardiogram (ECG) | Up to approximately 37 months
Part B: Number of participants with adverse events (AEs), immune-mediated adverse events (imAEs), adverse events of special interest (AESI), serious adverse events (SAEs) by Frequency | Up to approximately 37 months
Part B: Number of participants with adverse events (AEs), immune-mediated adverse events (imAEs), adverse events of special interest (AESI), serious adverse events (SAEs) by Severity | Up to approximately 37 months
Parts A and B: Change from Baseline in Eastern Cooperative Oncology Group Performance Scale (ECOG PS) score | Baseline and up to approximately 37 months
  ECOG PS is used for measuring how the disease impacts a participants daily living abilities. The grades for the scale range from 0 (fully active) to 5 (dead), with increasing severity.

CONTACTS AND LOCATIONS:
Locations (46):
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, CABA
  - GSK Investigational Site, Viedma
- Australia (2):
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Brazil (4):
  - GSK Investigational Site, Natal
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Copenhagen, Denmark
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
- France (3):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, München, Germany
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Pylaia Thessaloniki
  - GSK Investigational Site, Thessaloniki
- Japan (3):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, Oslo, Norway
- Panama (2):
  - GSK Investigational Site, Panama City
  - GSK Investigational Site, Punta Pacifica Panama City Panama
- Poland (2):
  - GSK Investigational Site, Józefów
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- GSK Investigational Site, Stockholm, Sweden
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
- United Kingdom (2):
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf